CLINICAL TRIAL: NCT06465914
Title: A Randomized, Double-blinded, Multicenter and Placebo-controlled Phase III Study to Evaluate the Efficacy, Immunogenicity and Safety of the 9-valent HPV Recombinant Vaccine (Hansenula Polymorpha) in Chinese Males Aged 18-45 Years
Brief Title: A Phase III Study to Evaluate the Efficacy, Immunogenicity and Safety of the 9-valent HPV Vaccine in Chinese Males
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9-HPV-3004
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Genital Wart; Penile Cancer; Anal Cancer; PIN-1; PIN2; PIN3; AIN1; AIN2; AIN3; HPV-Related Carcinoma
MeSH Terms: conditions — Condylomata Acuminata; Penile Neoplasms; Anus Neoplasms | interventions — Vaccines, Synthetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) vaccine (Experimental): Participants in this arm would receive 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine (Hansenula Polymorpha). Follow-up for the study encompassed Month 7 through Month 72.
  Interventions: Biological: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine (Hansenula Polymorpha)
- Placebo (Placebo Comparator): Participants in this arm would receive Placebo. Follow-up for the study encompassed Month 7 through Month 72.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine (Hansenula Polymorpha) — Subjects received 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule (0.5 mL intramuscular injection in the deltoid muscle).
  Arms: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) vaccine
Biological: Placebo — Subjects received 3 doses of Placebo according to a 0, 2, 6-month schedule (0.5 mL intramuscular injection in the deltoid muscle).
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the vaccine efficacy, immunogenicity and safety of the 9-valent (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Human Papillomavirus (HPV) Recombinant Vaccine (Hansenula Polymorpha) in Chinese male subjects aged 18-45 years. The primary hypothesis in the study is the 9-valent HPV recombinant vaccine reduces the incidence of vaccine HPV types-related genital warts compared with placebo in Chinese men.

DETAILED DESCRIPTION:
The primary aim of this clinical trial is to evaluate the efficacy of the 9-valent HPV vaccine in men aged 18-45 years old. It will also learn about the safety and immunogenicity of the 9-valent HPV vaccine.

Participants will inoculate the 9-valent HPV vaccine or a placebo according to the 0, 2, 6 month immunization program.

Visit the clinic on the 8th and 31st day after each dose of vaccination for the collection of safety information, keeping a diary of their symptoms and medications.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese men aged 18-45 years who can provide legal identification and have a sexual life history;
2. Subjects fully understands the study procedures, understands the risks and benefits associated with participating in the study, and voluntarily signs the informed consent;
3. Subjects are able to read, understand and fill in the research application forms such as diary CARDS and contact CARDS, and promise to participate in regular follow-up according to the study requirements;
4. Heterosexual men subjects must have exclusively female sexual partners and no more than 5 before enrollment;
5. MSM subject must have had sex with men within the past year (either insertive or receptive anal intercourse); and the cumulative number of sexual partners (including male and female sexual partners) does not exceed 5 before enrollment;
6. Subjects agree to provide effective contact information that can be used for communication with the researchers during the study;
7. Subjects consent to external anogenital lesion inspection and sample collection (including but not limited to wet swab collection and necessary biopsy) during the study period;
8. Subjects agree to take effective contraceptive measures from the first dose to 1 month after the last dose [male effective contraception including abstinence, male condom, vasectomy, etc.; female valid contraception including the pill (excluding emergency contraception), injection or embedded contraception, sustained-release topical contraceptives, hormonal patch, intrauterine devices (IUD), sterilization, diaphragm, cervical caps, etc.; safe period contraception, extracorporeal ejaculation, and emergency contraception are unacceptable contraception.]

Exclusion Criteria:

Initial inoculation exclusion criteria (If the "*" option is met during screening, the enrollment can be postponed and the re-screening can be rescheduled )

1. * Subjects with axillary temperature ≥37.3℃ 24 hours before the first vaccination;
2. * Higher blood pressure on the day of the first vaccination (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg);
3. * Sexual activity (including anal, vaginal/genital contact of the same or opposite sex) within 48 hours prior to the sampling visit; Self-shave hair from genital area within 24 hours prior to the genital examination visit (and/or using any post-shaving lotions or lubricants);
4. Have been or planned to be vaccinated with commercially available HPV vaccine; Have participated in or plan to participate in other HPV vaccine clinical trials;
5. Previous positive HPV test results (including types not included in the investigational vaccine) or related cytological abnormalities；
6. Previous or current HPV-related genital warts, penile/perianal/perineal intraepithelial neoplasia, penile/perianal/perineal cancer, anal intraepithelial neoplasia, or anal cancer;
7. Significant clinical evidence of external genital lesions and anal diseases (only MSM) suggesting the HPV infection during the external anogenital inspection before the first vaccination;
8. * Acute illness or acute episode of chronic disease, or use of antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days prior to vaccination;
9. * Received inactivated/recombinant/nucleic acid vaccine (non-attenuated vaccine) within 7 days prior to recruitment, or attenuated vaccine within 14 days prior to enrollment;
10. * Received any immune globulin or blood derived products within 3 months prior to enrollment, or plan to use any between the first vaccination and 1 month after full immunization;
11. * Received immunosuppressive therapy within 1 month prior to vaccination, such as immunosuppressive doses of glucocorticoids (dose reference: equivalent to prednisone 20mg/day for more than 7 days), or monoclonal antibodies, thymosin, interferon, etc., or plan to receive such treatment during the first dose until 1 month after full immunization, but topical administration (such as ointment, eye drops, inhalants or nasal sprays) is allowed;
12. Other investigational or unregistered products (drug or vaccine) that have been used within 3 months prior to the first dose or are planned to be used during the study period;
13. Present or have a history of convulsions (except febrile convulsions in childhood (0-14 years)), epilepsy, other serious neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.);
14. Present or have a history of mental illness or the family history;
15. There are contraindications to intramuscular injection, such as having been diagnosed with thrombocytopenia, any coagulation dysfunction, or being treated with anticoagulants;
16. Any condition resulting in asplenia or functional asplenia；
17. A history of severe allergic reactions requiring medical intervention (such as anaphylactic shock, anaphylactic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis (Arthus reaction), etc.); A history of severe adverse reactions to previous vaccination or a history of severe allergies (e.g. mouth and throat swelling, dyspnea, hypotension or shock, severe urticaria, etc.) to any vaccine component (histidine, sodium chloride, polysorbate 80, aluminum phosphate adjuvant and water for injection) ;
18. Subjects have been diagnosed with congenital or acquired immunodeficiency disease, such as: AIDS, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease or other immune disorders;
19. Currently have a serious infectious disease such as active tuberculosis, active viral hepatitis or acquired immunodeficiency syndrome (HIV infection);
20. Diagnosed with a serious congenital malformation or chronic disease that may interfere with the conduct or completion of the study, such as Down syndrome, heart disease, liver disease, kidney disease, diabetes with complications, or malignant tumors;
21. A history of drug abuse prior to enrolling, or a history of drug or alcohol abuse or dependence within the last year;
22. Subjects plan to permanently relocate from the region before the completion of the study or leave the region for a long period of time during the scheduled visit (affecting the scheduled visit time);
23. Investigators consider that the subjects have any condition that may interfere with the evaluation of the objectives of the study, or that participation in the study does not guarantee the maximum benefit of the subjects.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9000 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of genital wart | 0-72 month
  The incidence of histopathologic confirmed HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, 58-related genital wart in male subjects who are neutralizing antibody seronegative at day 0 and HPV-DNA negative from day 0 through 30-day after full immunization.

SECONDARY OUTCOMES:
The combined incidence of AIN1/2/3 and anal cancer in MSM | 0-72 month
  The combined incidence of histopathologic confirmed HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, 58-related AIN1/2/3 and anal cancer in MSM subjects who are neutralizing antibody seronegative at day 0 and HPV-DNA negative from day 0 through 30-day after full immunization.
The combined incidence of PIN1/2/3 and Penile/perianal/perineal cancer | 0-72 month
  The composite incidence of histopathologic confirmed HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, 58-related PIN1/2/3 and Penile/perianal/perineal cancer in male subjects who are neutralizing antibody seronegative at day 0 and HPV-DNA negative from day 0 through 30-day after full immunization.
The incidence of PI 12 | 0-72 month
  The incidence of 12-month persistent HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, 58-related infection detected from anogenital swabs, anal cells, or tissue samples which are successive sampled post Dose 3 immunization in subjects who are neutralizing antibody seronegative at day 0 and HPV-DNA negative from day 0 through 30-day after full immunization.
The incidence of PI 6 | 0-72 month
  The incidence of 6-month persistent HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, 58-related infection detected from anogenital swabs, anal cells, or tissue samples which are successive sampled post Dose 3 immunization in subjects who are neutralizing antibody seronegative at day 0 and HPV-DNA negative from day 0 through 30-day after full immunization.
The incidence of transient infection | 0-72 month
  The incidence of transient HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, 58-related infection detected from anogenital swabs, anal cells, or tissue samples which are successive sampled post Dose 3 immunization in subjects who are neutralizing antibody seronegative at day 0 and HPV-DNA negative from day 0 through 30-day after full immunization.
Immunogenicity | 0-72 month
  Immunogenicity: Geometric mean titer (GMTs) of HPV vaccine type-related neutralizing antibodies (pseudoviral neutralizing antibody assay) and lgG antibodies (ELISA assay) of subjects at day 0, 30-day after full immunization, 12, 36, and 72 months, and serological conversion rate (SCR) was calculated.
The incidence of solicited adverse events | 0-7 days after each dose of vaccine
  The incidence of solicited adverse events within 30 minutes and 0-7 days after each dose of vaccine for all subjects;
The incidence of unsolicited adverse events | 0-30 days after each dose of vaccine
  The incidence of unsolicited adverse events within 0-30 days after each dose of vaccine for all subjects;
The incidence of serious adverse events | 0-72 month
  The incidence of all serious adverse events that occurred between the first dose and the last follow-up in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Lidong Gao, Master, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention; Long Sui, Doctor, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (5):
- China (5):
  - Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi
  - Hunan Center for Disease Control and Prevention, Changsha, Hunan
  - Shanxi Provincial Disease for Control and Prevention, Taiyuan, Shanxi
  - Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan
  - Yunnan Center for Disease Control and Prevention, Kunming, Yunnan